CLINICAL TRIAL: NCT03309735
Title: Multicenter Open Prospective Comparative Non-interventional Study of Therapy for Threatened Miscarriage With Medicinal Products Utrogestan, 200 mg Capsules (Besins Healthcare SA, Belgium), and Duphaston, 10 mg Coated Tablets (Abbott Healthcare Products B.V., the Netherlands)
Brief Title: Non-interventional Study of Therapy for Threatened Miscarriage
Status: Completed | Type: Observational
Sponsor: Besins Healthcare (Industry)
Collaborators: Clinical Research Laboratory, CRO, Russia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0717-1
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Threatened Miscarriage
Keywords: threatened miscarriage; miscarriage; micronized progesterone; dydrogesterone
MeSH Terms: conditions — Abortion, Threatened; Abortion, Spontaneous | interventions — Progesterone; Utrogestan; Dydrogesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Utrogestan, 200 mg orally thrice a day until acute symptoms of the threat of termination of pregnancy (scarlet discharge from the genital tract, pain in the abdomen) and then Utrogestan vaginally 200 mg twice a day and 200 mg orally once a day before bed
  Interventions: Drug: Micronized progesterone
- 2: Utrogestan vaginally 200 mg twice a day and 200 mg orally once a day before bed
  Interventions: Drug: Micronized progesterone
- 3: Duphaston, orally 40 mg once, then 10 mg every 8 hours until the symptoms disappear
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Micronized progesterone — Utrogestan, 200 mg orally thrice a day until acute symptoms of the threat of termination of pregnancy (scarlet discharge from the genital tract, pain in the abdomen) and then Utrogestan vaginally 200 mg twice a day and 200 mg orally once a day before bed
  Other Names: Utrogestan
  Groups: 1
Drug: Micronized progesterone — Utrogestan vaginally 200 mg twice a day and 200 mg orally once a day before bed
  Other Names: Utrogestan
  Groups: 2
Drug: Dydrogesterone — Duphaston, orally 40 mg once, then 10 mg every 8 hours until the symptoms disappear
  Other Names: Duphaston
  Groups: 3

SUMMARY:
Study the efficacy and safety of therapy for threatened miscarriage with medicinal products Utrogestan (micronized progesterone), 200 mg capsules (Besins Healthcare SA, Belgium), and Duphaston (Dydrogesterone), 10 mg coated tablets (Abbott Healthcare Products B.V., the Netherlands)

DETAILED DESCRIPTION:
Open comparative non-interventional study.

During the study three visits are planned:

Visit 1 (enrollment) is conducted when the patient is hospitalized in a hospital (providing medical care to pregnant women diagnosed with threatened miscarriage) due to the threat of miscarriage when the inclusion/exclusion criteria are met (women aged 18-35 years with a confirmed threat of miscarriage with a gestation period of 8 to 22 full weeks). Depending on the chosen therapy tactics (this therapy is routine in Russia), all patients are allocated to one of the three study groups:

Group I receives Utrogestan (micronized progesterone), 200 mg orally thrice a day until acute symptoms of the threat of termination of pregnancy (scarlet discharge from the genital tract, pain in the abdomen) and then Utrogestan vaginally 200 mg twice a day and 200 mg orally once a day before bed; Group II receives Utrogestan (micronized progesterone) vaginally 200 mg twice a day and 200 mg orally once a day before bed; Group III receives Duphaston (Dydrogesterone), orally 40 mg once, then 10 mg every 8 hours until the symptoms disappear.

Visit 2 (on the third day of the study/hospitalization). If pregnancy is interrupted earlier, Visit 3 is made.

Visit 3 (on the day of discharge from the hospital: with prolonged or interrupted pregnancy)

Routine clinical procedures (accepted in Russia) will be performed during the study:

* Collection of demographic and anthropometric data (age, height, body weight);
* Collection of complaints, medical and obstetric-gynecological history;
* Measurement of blood pressure, heart rate, respiratory rate and body temperature;
* Gynecological examination with the help of gynecological specula;
* Vaginal bimanual examination;
* Transvaginal ultrasound, determination of viability of uterine pregnancy (determination of embryo/fetal heartbeat);
* Assessment of the severity of the patient's condition according to Clinical Global Impression scale;
* Evaluation of psycho-emotional status dynamically using Zigmond-Snaith Hospital Anxiety and Depression Scale;

Efficacy will be evaluated using primary and secondary efficacy endpoints.

Primary efficacy endpoint:

• Discharge from the hospital with prolonged pregnancy;

Secondary efficacy endpoint:

* Speed of arrest of symptoms of threatened miscarriage (blood discharge from the genital tract and drawing pains in the lower abdomen);
* Duration of hospitalization;
* Severity of patient's condition dynamically in the course of therapy;
* Psycho-emotional status of women dynamically in the course of therapy;

Criteria for safety evaluation:

• Evaluation of AE/SAE. All adverse events (As) and serious adverse events (SAE) will be recorded, starting from the moment of signing of informed consent before the end of participation in the study (before discharge from the hospital).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent of the patient to participate in the study;
* Women aged 18-35 years;
* Progressive uterine pregnancy at the time of inclusion in the study from 8 to 22 full weeks;
* Drawing pains in the lower abdomen, lumbar region;
* Scanty blood discharge from the genital tract;
* Palpitation of the fetus revealed by ultrasound;
* Prescription by attending physician of Utrogestan or Duphaston, depending on chosen treatment tactics.

A physician should decide on the therapy, as well as tactics of further management of pregnancy before the patient is enrolled in the study and regardless of it.

Exclusion Criteria:

* Stimulated ovulation, use of assisted reproductive technologies;
* Abnormalities in the structure of the uterus;
* Amputation of the cervix;
* Uterine myoma with submucosal location of the node (a clinically significant size);
* Karyotype anomalies of parents (if applicable);
* Aneuploidy, anembrion, fetal malformations, as established causes of loss of previous pregnancies;
* Congenital thrombophilia: factor V gene mutation (Leiden mutation), mutation of the prothrombin gene (if applicable);
* Non-developing pregnancy;
* Other clinically significant causes of miscarriage identified during examination (including but not limited to): pre-pregnancy diabetes, pre-pregnancy uncompensated thyroid dysfunction, history of malignant tumors or current tumors, psychiatric illnesses;
* STDs at the time of inclusion in the study;
* Administration of enzyme-inducing medicinal products (anticonvulsants, antipsychotics, antidepressants, tranquilizers), use of psychoactive substances before and during pregnancy;
* Multiple pregnancy;
* Patients previously included in this study, but who withdrew from the study for any reason;
* Contraindications to therapy with Utrogestan and Duphaston, listed in approved prescribing instructions;
* Contraindications to pregnancy prolongation;
* Any other clinical conditions that, as seen by investigator, contradict inclusion criteria, may lead to the early termination of the patient's participation in the study or make it difficult to interpret the results of the latter;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18-35 years with a confirmed threat of miscarriage with a gestation period of 8 to 22 full weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1241 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Prolongation of pregnancy | Through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  Discharge from the hospital with prolonged pregnancy

SECONDARY OUTCOMES:
Speed of arrest of acute symptoms of threatened miscarriage | Through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  Speed of arrest of symptoms of threatened miscarriage (blood discharge from the genital tract and drawing pains in the lower abdomen)
Duration of hospitalization | Through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  Duration of hospitalization
Severity of patient's condition | Through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  Severity of patient's condition dynamically in the course of therapy
Psycho-emotional status of patients | Through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  Psycho-emotional status of women dynamically in the course of therapy

OTHER OUTCOMES:
Evaluation of AE/SAE | From the moment of signing of informed consent through study completion (until the date of patient discharge from hospital, an averade 7-14 days)
  All adverse events (AE) and serious adverse events (SAE) will be recorded during the study

CONTACTS AND LOCATIONS:
Overall Officials: Igor Manuhin, PhD, Principal Investigator — Moscow State University of Medicine and Dentistry named after A.I. Evdokimov
Locations (17):
- Russia (17):
  - City Clinical Hospital of the Demsk District, Ufa, Bashkortostan Republic
  - Maternity hospital №1, Krasnoyarsk, Krasnoyarsk Region
  - Regional perinatal center, Kursk, Kursk Oblast
  - Chekhov district hospital №1, Chekhov, Moscow Oblast
  - Central district hospital, Zhukovsky, Moscow Oblast
  - Center for Family Planning and Reproduction, Novosibirsk, Novosibirsk Oblast
  - Maternity hospital №2, Omsk, Omsk Oblast
  - Maternity hospital №6, Omsk, Omsk Oblast
  - Сity hospital №7, Samara, Samara Oblast
  - Stavropol Central District Hospital, Stavropol, Stavropol Kray
  - Сentral city hospital, Kamensk-Uralsky, Sverdlovsk Oblast
  - City Clinical Hospital №16, Kazan', Tatarstan Republic
  - City Clinical Hospital № 8, Voronezh, Voronezh Oblast
  - Regional Perinatal Center, Yaroslavl, Yaroslavl Oblast
  - City Clinical Hospital №68, Moscow
  - Pirogov Russian National Research Medical University (RNRMU), Moscow
  - Maternity hospital №17, Moscow

IPD SHARING:
Plan to Share IPD: No